CLINICAL TRIAL: NCT03646383
Title: Study of the Feasibility of Radiofrequency Ablation of Benign Thyroid Nodules by Percutaneous Radiological Approach
Brief Title: Study of the Feasibility of Radiofrequency Ablation of Benign Thyroid Nodules
Acronym: TRAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/17/0352; 2018-A00669-46 (Other: ID-RCB)
Record Dates: First submitted 2018-03-25; First posted 2018-08-24 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Benign Thyroid Nodules
Keywords: benign thyroid nodule; radiofrequency; symptomatic thyroid nodule
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with radiofrequency (Experimental): Treatment of symptomatic benign nodules with radiofrequency ablation as an alternative to surgical treatment
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — The procedure will include an ultrasound with radiofrequency ablation of the benign thyroid nodule percutaneously

SUMMARY:
The purpose of the present protocol is to evaluate the response rate to treatment of these symptomatic benign nodules with radiofrequency as an alternative to surgical treatment.

This thyroid nodules ablation with radiofrequency will be directed by a single percutaneous procedure guided by ultrasound. The procedure includes an ultrasound with percutaneously radiofrequency ablation of benign thyroid nodule. Clinical and ultrasonographic monitoring will last a year with consultations at 2 weeks (consultation only), 3 months, 6 months and 1 year (consultation, ultrasound TSH). The success of this procedure will be controlled with 3 successive ultrasounds the following year. The expected results are a decrease in the size of the nodule by at least 50% and a reduction in the functional and aesthetic discomfort, with less frequent complication than what is expected with surgery. The present study also intends to determine the medico economic impact of this technique compared to surgery.

DETAILED DESCRIPTION:
Thyroid benign nodules represent a major public health problem because they are very common (subclinical nodules were found in half of woman beyond 60 years). The main risk factors include age, female gender, parity, smoking and family history of thyroid nodules or thyroiditis. The assessment is based on biology, ultrasound and fine needle aspiration and intends to determine the benign nature (95%) or cancer (5%) of the nodules and if they are functional or not (toxic nodule). Most benign nodules are asymptomatic but some of them because of their size and location can cause a functional disorder (compression or swallowing disorder) or aesthetic and psychological resounding.In current practice, these nodules are sometimes treated with surgery that impact on patient quality of life (need to take L-Thyroxine, difficulties related to the possible occurrence of complications like hypoparathyroidism or laryngeal paralysis) and socio-economic constraints especially when complications occur. To limit the number of unnecessary and potentially risky surgeries, patients should therefore be well selected. If surgery is the preferred treatment of thyroid cancer, alternative techniques like radiofrequency seem interesting for benign nodules.

ELIGIBILITY:
Inclusion Criteria:

* Euthyroid or hypothyroidism properly substituted with normal TSH
* Benin nodule proved by FNA (Bethesda) and normal Calcitonin
* Nodule size> 1cm and / or increase in size
* Single nodule or asymptomatic nodules associated
* Symptomatic nodule with functional impairment and / or aesthetic Patient Agreement
* Patient with insurance coverage
* Written agreement for participation

Exclusion Criteria:

The exclusion criteria are related to the histological nature of the nodule and the necessary of the procedure:

* Allergy to local anesthetics
* FNA non-contributory or suspicious nodule (Bethesda)
* Multiple nodules more than 2cm
* Hyperthyroidism or hyperparathyroidism associated requiring surgical intervention.
* Taking a treatment with anticoagulant or double antiplatelet
* Patient with a Pacemaker
* Contralateral laryngeal paralysis in nodule
* Purely cystic nodule
* Nodule in contact with the recurrent nerve
* Patient Refusal
* Pregnant and breastfeeding women
* Patient trust, guardianship or safeguard justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Procedure response rate | 6 months
  First estimate of the procedure response rate (patient with complete procedure in percentage)

SECONDARY OUTCOMES:
Change in nodular volume | at 6 and 12 months
  compared to the volume measured at inclusion. This reduction will be estimated in absolute value and in relative value (percentage reduction for a given subject)
volume change of nodules by at least 50 percent, at 6 months | at 6 months
  Percentage of patients with a volume decrease of at least 50 percent, 6 months after the procedure. Patients for which the procedure could not be fully performed will be counted among patients who have not had a reduction of at least 50 percent
volume change of nodules by at least 50 percent, at 12 months | at 12 months
  Percentage of patients with a volume decrease of at least 50 percent, 12 months after the procedure. Patients for which the procedure could not be fully performed will be counted among patients who have not had a reduction of at least 50 percent
complete disappearance of symptoms | at 12 months
  The symptoms will be evaluated by a visual analogue scale of 0 to 10 as proposed by the Korean consensus. The symptoms assessed will be: cervical pain, dysphagia, foreign body sensation, discomfort, coughing.
aesthetic change | at 3, 6 and 12 months
  This improvement will be evaluated with a 4-level scale (no clinically detectable nodule 0, palpable nodule 1, visible nodule on swallowing 2, spontaneously visible nodule 3) as proposed by the Korean consensus. The improvement will be defined by the transition to the lower category.
one or more complications | at 6 and 12 months
  In particular, the following will be investigated: signs of cutaneous involvement such as burns, hematoma and intra-nodular bleeding, recurrent paralysis, superinfections, tracheal or esophageal wounds.
Assessment of pain during the procedure with visual analogue scale | between Day 1 and Day 15
  Evaluation of the pain during the procedure using a visual analogue scale from 0 to 10 established at the end of the procedure
patients requiring L-thyroxine replacement therapy | at 6 and 12 months
  Percentage of patients requiring L-thyroxine replacement therapy
Economic evaluation from the point of view of the hospital | Between Day 1 and 12 months
  evaluation, from the point of view of the hospital, of the production cost of the new technique
patients who have used analgesics | between Day 1 and Day 15
  Percentage of patients who have used analgesics during and after the procedure
Economic evaluation from the point of view of the health insurance | Between Day 1 and 12 months
  Evaluation, from the point of view of health insurance, of the cost of the care of patients who benefited from the new technique

CONTACTS AND LOCATIONS:
Overall Officials: Claire RENAUD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Hôpital Larrey, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967
- [Background] Fuller CW, Nguyen SA, Lohia S, Gillespie MB. Radiofrequency ablation for treatment of benign thyroid nodules: systematic review. Laryngoscope. 2014 Jan;124(1):346-53. doi: 10.1002/lary.24406. Epub 2013 Oct 22. PMID 24122763
- [Background] Deandrea M, Sung JY, Limone P, Mormile A, Garino F, Ragazzoni F, Kim KS, Lee D, Baek JH. Efficacy and Safety of Radiofrequency Ablation Versus Observation for Nonfunctioning Benign Thyroid Nodules: A Randomized Controlled International Collaborative Trial. Thyroid. 2015 Aug;25(8):890-6. doi: 10.1089/thy.2015.0133. Epub 2015 Jul 13. PMID 26061686
- [Background] Hong MJ, Na DG, Baek JH, Sung JY, Kim JH. Cytology-Ultrasonography Risk-Stratification Scoring System Based on Fine-Needle Aspiration Cytology and the Korean-Thyroid Imaging Reporting and Data System. Thyroid. 2017 Jul;27(7):953-959. doi: 10.1089/thy.2016.0603. Epub 2017 May 19. PMID 28463597
- [Background] Chen F, Tian G, Kong D, Zhong L, Jiang T. Radiofrequency ablation for treatment of benign thyroid nodules: A PRISMA-compliant systematic review and meta-analysis of outcomes. Medicine (Baltimore). 2016 Aug;95(34):e4659. doi: 10.1097/MD.0000000000004659. PMID 27559968